CLINICAL TRIAL: NCT03767829
Title: A Phase 1/2, Randomized, Double-blind, Placebo-controlled, Single-ascending and Multiple-dose, Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics Study of Subcutaneously Administered ALN-AAT02 in Healthy Adult Subjects and Patients With ZZ Type Alpha-1 Antitrypsin Deficiency Liver Disease
Brief Title: A Study of ALN-AAT02 in Healthy Participants and Participants With ZZ Type Alpha-1 Antitrypsin Deficiency Liver Disease
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The sponsor decided not to proceed with Part B for business reasons.
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALN-AAT02-001; 2018-001362-41 (EudraCT Number)
Record Dates: First submitted 2018-12-05; First posted 2018-12-07 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: ZZ Type Alpha-1 Antitrypsin Deficiency Liver Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part A: SAD: ALN-AAT02 (Experimental): Participants will be administered a single dose of ALN-AAT02.
  Interventions: Drug: ALN-AAT02
- Part A: SAD: Placebo (Placebo Comparator): Participants will be administered a single dose of matching placebo.
  Interventions: Drug: Placebo
- Part B: MAD: ALN-AAT02 (Experimental): Participants will be administered multiple doses of ALN-AAT02.
  Interventions: Drug: ALN-AAT02
- Part B: MAD: Placebo (Placebo Comparator): Participants will be administered multiple doses of matching placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALN-AAT02 — ALN-AAT02 will be administered subcutaneously (SC) at dose levels planned for Part A.
  Arms: Part A: SAD: ALN-AAT02
Drug: Placebo — Sterile normal saline (0.9% NaCl) matching volume of ALN-AAT02 doses will be administered SC.
  Arms: Part A: SAD: Placebo; Part B: MAD: Placebo
Drug: ALN-AAT02 — ALN-AAT02 will be administered subcutaneously (SC). Part B dose levels to be determined upon review of data from Part A.
  Arms: Part B: MAD: ALN-AAT02

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of single or multiple doses of ALN-AAT02. The study will be conducted in 2 sequential phases in which Part A will be a single-ascending dose (SAD) phase in healthy participants, and Part B will be a multiple-ascending dose (MAD) phase in participants with ZZ type alpha-1 antitrypsin deficiency (PiZZ) and biopsy-proven alpha-1 antitrypsin (AAT) deficiency-associated liver disease.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 to 65 years, inclusive;
* Has normal 12-lead electrocardiogram (ECG);
* Has body mass index (BMI) between 18 and 30 kg/m^2, inclusive;
* Has been a nonsmoker for at least 5 years before screening;
* Part A only: Has Alpha-1 antitrypsin (AAT) levels within normal limits;
* Part A only: Has adequate Forced Expiratory Volume in 1 second (FEV1) and adequate FEV1/forced vital capacity ratio;
* Part B only: Has documented ZZ type AAT by genotype;
* Part B only: Has liver biopsy within 90 days of the first dose of study drug demonstrating ZZ type alpha-1 antitrypsin deficiency (PiZZ AATD) liver disease;
* Part B only: Has adequate post-bronchodilator FEV1 and adequate diffusing capacity of the lung for carbon monoxide;
* Part B only: If on any maintenance medication, is likely to be able to remain on a stable medication regimen for the duration of the study (no new medications within 30 days prior to first dose of study drug).

Exclusion Criteria:

* Has known human immunodeficiency virus (HIV), hepatitis C virus (HCV) or hepatitis B virus (HBV) infection;
* Has clinically significant abnormal laboratory results;
* Received an experimental drug within 30 days of dosing;
* Has a history of multiple drug allergies or history of allergic reaction to an oligonucleotide or N-acetylgalactosamine (GalNAc);
* Part A only: Has estimated glomerular filtration equal to or below 60 mL/min/1.73 m^2 at screening;
* Part A only: Has a history of asthma or recurrent or chronic lung disease, excluding resolved childhood asthma;
* Part A only: Has a history of chronic liver disease;
* Part B only: Has estimated glomerular filtration equal to or below 45 mL/min/1.73 m^2 at screening;
* Part B only: Received an augmentation therapy for AAT deficiency within 8 weeks of first dose of study drug;
* Part B only: Has a history of chronic liver disease from any known cause other than ZZ type AAT deficiency;
* Part B only: Has a history of hepatic encephalopathy;
* Part B only: Has a history of gastrointestinal bleeding or ascites.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2020-06-25 (Actual); Study Completion 2020-06-25 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Treatment Emergent Adverse Events (TEAEs) | Part A: up to approximately 12 months; Part B: up to approximately 18 months

SECONDARY OUTCOMES:
Change From Baseline in Serum Levels of Alpha-1 Antitrypsin (AAT) | Part A: baseline up to Day 85 and every 84 days up to approximately 12 months; Part B: baseline up to Day 169 and every 84 days up to approximately 18 months
Maximum Observed Plasma Concentration (Cmax) for ALN-AAT02 | Part A: Days 1, 2, 3, 8 and 15; Part B: Days 1, 2, 3, 29, 85, 86 and 87
Time to Reach Cmax (tmax) for ALN-AAT02 | Part A: Days 1, 2, 3, 8 and 15; Part B: Days 1, 2, 3, 29, 85, 86 and 87
Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) for ALN-AAT02 | Part A: Days 1, 2, 3, 8 and 15; Part B: Days 1, 2, 3, 29, 85, 86 and 87
Apparent Terminal Elimination Half-life (t1/2) for ALN-AAT02 | Part A: Days 1, 2, 3, 8 and 15; Part B: Days 1, 2, 3, 29, 85, 86 and 87
Fraction Eliminated in Urine (fe) of ALN-AAT02 | Part A: Day 1; Part B: Days 1 and 85
Amount of Full Length Drug Excreted in Urine (Ae) of ALN-AAT02 | Part A: Day 1; Part B: Days 1 and 85

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Alnylam Pharmaceuticals
Locations (1):
- Clinical Trial Site, London, United Kingdom